CLINICAL TRIAL: NCT03101956
Title: Spinal Manipulation for Improving Hip and Knee Muscle Strength in Patients With Patellofemoral Pain Syndrome - A Randomized, Placebo-Controlled, Clinical Trial
Brief Title: Lumbar Manipulation for Hip and Muscle Strength
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16-01718
Record Dates: First submitted 2017-03-30; First posted 2017-04-05 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-11

CONDITIONS: Patellofemoral Pain Syndrome; Anterior Knee Pain Syndrome
Keywords: Spine Manipulation
MeSH Terms: conditions — Patellofemoral Pain Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- L/S Manipulation Study Group (Experimental)
  Interventions: Procedure: Lumbar Spine Manipulation
- Control Group (Active Comparator)
  Interventions: Procedure: Lumbar Spine Manipulation Placebo

INTERVENTIONS:
Procedure: Lumbar Spine Manipulation — • The subject will be placed in sidelying on a treatment table. Facing the subject, the therapist will position the subject's superior thigh in flexion and rotate the subject's upper trunk to the opposite side. The therapist will place his cephalad forearm along the subject's superior lateral trunk and the caudal forearm along the subject's iliac crest and lateral hip. Lastly, the therapist will roll the subject towards himself or herself.
  Other Names: Sidelying lumbosacral thrust joint manipulation
  Arms: L/S Manipulation Study Group
Procedure: Lumbar Spine Manipulation Placebo — The subject will be placed in sidelying on a treatment table. Facing the subject, the therapist will position both hips and knees in approximately 45° of flexion. The therapist will place his or her cephalad forearm along the subject's superior lateral trunk and the caudal forearm along the subject's iliac crest and lateral hip. Lastly, the therapist will roll the subject towards himself or herself.
  Other Names: Sidelying lumbosacral thrust joint manipulation placebo
  Arms: Control Group

SUMMARY:
The aim of this double blind, randomized, placebo-controlled clinical trial is to investigate the immediate effects of spinal manipulation on hip and knee muscle strength and pain-free deep squat range of motion in order to answer several conceptual and practical research questions

DETAILED DESCRIPTION:
This prospective, double-blind, randomized control trial clinical will use a multigroup pretest-posttest control design with 1 treatment arm and 1 control arm. Interpreted within the biopsychosocial model and the International Classification of Functioning, Disability and Health (ICF) framework, this research will measure the outcomes between patellofemoral pain syndrome (PFPS), the health condition, and contextual factors, particularly personal factors. It will address personal factors such as gender and age but will not address environmental factors. This research includes tests and measures of two of the three levels of human functioning, or domains, impairments to body functions and structures and activity limitations. Muscle strength testing is an impairment-level measure and pain-free deep squat range of morion (ROM) is an activity limitation-level measure.

ELIGIBILITY:
Inclusion Criteria:

* Referred to out-patient physical therapy for a knee condition and a chief complaint of anterior knee pain
* Anterior knee pain with squatting
* Agreed to be in the study and signed the informed consent document

Exclusion Criteria:

* Presence of any medical 'red flags' suggestive of pain that is not of musculoskeletal origin
* Osteoporosis or recent fracture of the hip or spinal joints
* Spinal or hip joint surgery or prosthesis
* Knee surgery on the affected knee within the last 6 months
* Spinal instability (Grade II spondylolithesis or greater), spondyloarthritides, or severe spinal misalignment
* Nervous system disease or disorder
* Pregnant
* Lumbar nerve root compression (any of the following signs present)
* Positive straight leg raise (SLR) test less than 45°
* Marked paresis involving a major muscle group of the lower extremity
* Diminished, and asymmetric (lower than uninvolved side), lower extremity
* muscle stretch reflex
* Diminished or absent sensation to pinprick in any lower extremity dermatome

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2019-06-21 (Actual); Study Completion 2019-06-21 (Actual)

PRIMARY OUTCOMES:
Muscle Strength using dynamometer | 1 Day
  Hand-held dynamometry involves the use of a dynamometer that is held by a tester and applied to the tested segment of a patient's body.
Score on European Quality of Life-5 Dimensions Questionnaire (EQ-5D) | 1 Day
  The EQ-5D-3L descriptive system comprises the following 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, extreme problems

SECONDARY OUTCOMES:
Subject's report of pain on the Numeric Pain Rating Scale (NPRS) at rest | 1 Day
  Numeric Pain Rating Scale

CONTACTS AND LOCATIONS:
Overall Officials: Michael D'Agati, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States